CLINICAL TRIAL: NCT05690113
Title: Translation and Validation in French of a Child Psychotrauma Identification Scale - the CATS (Child and Adolescent Trauma Screen)
Brief Title: Translation and Validation of the "Children and Adolescent Trauma Screen" in French
Acronym: French-CATS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0390; 2022-A02018-35_22 (Other: ANSM)
Record Dates: First submitted 2022-11-29; First posted 2023-01-19 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Child Psychiatry; Adolescent Psychiatry
Keywords: psychotraumatism; children; adolescent; scale; french translation; validation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical population: 250 children aged from 7 to 17 will be recruited in 6 clinical departments (child and adolescent psychiatry, forensic medicine, psychotraumatism centers) They will complete the CATS scale as well as the SCARED (Screen for Child Anxiety and Related Disorders). Their parents will also complete the CATS and the SDQ (Strength and Difficulties Questionnaire) to assess convergent and divergent validity.
  Interventions: Procedure: CATS scale
- Non-clinical population: 250 children aged from 7 to 17 will be recruited in schools They will complete the CATS scale as well as the SCARED (Screen for Child Anxiety and Related Disorders). Their parents will also complete the CATS and the SDQ (Strength and Difficulties Questionnaire) to assess convergent and divergent validity.
  Interventions: Procedure: CATS scale

INTERVENTIONS:
Procedure: CATS scale — During the inclusion visit (J0), enrolled children will complete the CATS scale as well as the SCARED (Screen for Child Anxiety and Related Disorders). Their parents will also complete the CATS and the SDQ (Strength and Difficulties Questionnaire).
  Other Names: SCARED scale; SDQ scale

SUMMARY:
Child psychotraumatism and complex psychotraumatism, mainly consecutive to child maltreatment, is a major unaddressed public health issue.

The investigators aim to translate and validate a screening scale to help professionals to better detect and refer children at risk of psychotraumatism.

This study aims to validate the psychometric properties of a french version of the CATS 2.0, in partnership with the original authors of the scale.

ELIGIBILITY:
Inclusion Criteria:

* child aged between 7 and 17
* at least an adult of reference (parent or tutor) reachable
* agreement of adult of reference
* for clinical population : have been potentially exposed to a potential traumatic event (according to DSM-V)

Exclusion Criteria:

* non-mastery of French language

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study will focus on children and adolescents between 7 and 17 years who have been potentially exposed to a traumatic event and who are treated in one of the participating services.
  This study will also focus on children and adolescents aged 7 to 17 years in the general population, enrolled in school in the Grenoble Academy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2024-03-09 (Actual); Study Completion 2024-03-09 (Actual)

PRIMARY OUTCOMES:
Psychometric properties of the Children and Adolescent Trauma Screen (CATS) scale | Day 0 (D0)
  Construct validity (structural validity, convergent-divergent validity), intraclass correlation coefficients, and internal consistency analysis will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Pauline ESPI, MD, Principal Investigator — Centre Régional de Psychotraumatisme, Hôpital Edouard Herriot, Hospices Civils de Lyon
Locations (6):
- France (6):
  - Service de Psychopathologie de l'Enfant et l'Adolescent, Hôpital Femme Mère Enfant, Bron
  - Laboratoire de Psychologie et de NeuroCognition, Domaine Universitaire de Jacob Bellecombette, Chambéry
  - Centre Régional de Psychotraumatisme, Hôpital Edouard Herriot, Lyon
  - Service de Médecine Légale, Hôpital Edouard Herriot, Lyon
  - Centre d'Evaluation de Psychotraumatisme Pédiatrique, CHU Lenval, Nice
  - Centre Psychotrauma Grand Est Alsace Nord, Hôpital civil et hôpital de l'Elsau, Strasbourg